CLINICAL TRIAL: NCT01886573
Title: Genome-Wide Methylation and Gene Re-expression Analysis of Resectable Lung Tumor Tissue Pairs Obtained Pre- and Post-Treatment With 5-Azacytidine and Entinostat
Brief Title: Azacitidine and Entinostat in Treating Patients With Newly Diagnosed Stage IA-IIIA Non-Small Lung Cancer Undergoing Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01186; NCI-2013-01186 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CTEP 9431; INST 1117 (Other: University of New Mexico); 9431 (Other: CTEP); P30CA118100 (NIH); R21CA161561 (NIH)
Record Dates: First submitted 2013-06-21; First posted 2013-06-26 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Stage IA Non-Small Cell Lung Carcinoma; Stage IB Non-Small Cell Lung Carcinoma; Stage IIA Non-Small Cell Lung Carcinoma; Stage IIB Non-Small Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Azacitidine; entinostat

ARMS (1):
- Treatment (azacitidine, entinostat) (Experimental): Patients receive azacitidine SC on days 1-6 and 8-10 and entinostat PO on days 3 and 10. Patients undergo surgery between days 11-20 (this period can be extended 10 more days if adverse events from therapy impose a surgical risk).
  Interventions: Drug: Azacitidine; Drug: Entinostat; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Azacitidine — Given SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; MS 27-275; MS-275; SNDX-275
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This pilot clinical trials studies azacitidine and entinostat in treating patients with newly diagnosed stage IA-IIIIA non-small cell lung undergoing surgery. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Entinostat may stop the growth of cancer tumor cells by blocking some of the enzymes needed for cell growth. Giving azacitidine with entinostat may be an effective treatment for non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To measure reversal of aberrant genome-wide promoter methylation and gene re-expression in paired, pre- and post- treatment lung tumor tissue pairs from patients with newly diagnosed, surgically resectable non-small cell lung cancer before and after exposure to a single neoadjuvant cycle of 5-azacytidine (azacitidine) and entinostat.

SECONDARY OBJECTIVES:

I. To measure the 3-year disease-free survival of operable non-small cell lung cancer (NSCLC) patients who receive 1 cycle of preoperative epigenetic treatment.

II. To determine any potential toxicities, and reversibility of toxicities, of a single pre-operative cycle of 5-azacytidine and entinostat.

OUTLINE:

Patients receive azacitidine subcutaneously (SC) on days 1-6 and 8-10 and entinostat orally (PO) on days 3 and 10. Patients undergo surgery between days 11-20 (this period can be extended 10 more days if adverse events from therapy impose a surgical risk).

After completion of study treatment, patients are followed up at 4 weeks, every 3 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a diagnostic biopsy, including computed tomography (CT)-guided or bronchoscopic for suspected diagnosis of NSCLC
* Able to understand and sign an informed consent discussing the risks and benefits of obtaining a concurrent research biopsy; patients who have a fresh frozen biopsy available secondary to institutional tissue collection protocols may substitute such a biopsy for the study-required pre-treatment biopsy
* Histologically confirmed diagnosis of operable NSCLC that has not been previously treated
* Clinical stage IA-IIIA
* Appropriate candidate for surgical management, in the opinion of the treating thoracic surgeon
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 at the time of initiation of neoadjuvant epigenetic therapy
* Absolute neutrophil count > 1,000/mcL
* Platelets > 100,000/mcL
* Total bilirubin < 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x institutional ULN
* Creatinine < 1.5 x institutional ULN
* Able to understand and sign an informed consent
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Inclusion of women and minorities:

  * Both men and women and members of all races and ethnic groups are eligible for this trial; the coordinating center will be responsible for ensuring each participating site is accruing a representative sample consistent with the estimate of population representation in the site's geographical location for race and ethnic groups as determined by the Census Bureau to assure overall target goals are met

Exclusion Criteria:

* Patients who have received prior chemotherapy or radiation for their diagnosis of lung cancer
* Patients may not be receiving any other investigational agent
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to entinostat or 5-azacytidine
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated on this protocol
* Any co-morbid condition that' in the view of the attending physician' renders the patient at high risk from treatment complications
* Human immunodeficiency virus (HIV) positive patients on combination antiretroviral therapy are ineligible
* Known or suspected hypersensitivity to azacitidine or mannitol
* Patients with advanced malignant hepatic tumors
* Use of anti-neoplastic or anti-tumor agents that are not part of the study therapy, including chemotherapy, radiation therapy, immunotherapy, and hormonal anticancer therapy, is not permitted while participating in this study; Note: study participants with stage II or III NSCLC, or stage I NSCLC with tumor size greater than 4 cm, should be offered standard adjuvant platinum-based chemotherapy in accordance with local practice (post-operatively)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in aberrant genome-wide promoter methylation | Baseline up to day 20
  Genome-wide DNA methylation and gene expression profiles of each pre- and post-treatment tumor will be assessed using validated DNA methylation and gene expression arrays. Response will be measured based on the degree of epigenomic reprogramming (i.e., number of genes affected, degree of demethylation, and class of genes [e.g., PRC2]) and pathways affected.
Change in gene expression | Baseline up to day 20
  Genome-wide DNA methylation and gene expression profiles of each pre- and post-treatment tumor will be assessed using validated DNA methylation and gene expression arrays. Response will be measured based on the degree of epigenomic reprogramming (i.e., number of genes affected, degree of demethylation, and class of genes [e.g., PRC2]) and pathways affected.

SECONDARY OUTCOMES:
Disease-free survival | Up to 3 years
Reversibility of toxicities | Up to 4 weeks after surgery
Toxicities, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.02 | Up to 4 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Montaser Shaheen, Principal Investigator — University of New Mexico
Locations (3):
- United States (3):
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - University of New Mexico, Albuquerque, New Mexico
  - University of Texas Southwestern Medical Center, Dallas, Texas